CLINICAL TRIAL: NCT01321931
Title: Multiple-dose Nicotine Pharmacokinetics With Three Oral Nicotine Replacement Products. A Study in Healthy Smokers.
Brief Title: Multiple-dose Nicotine Pharmacokinetics With Three Oral Nicotine Replacement Products
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NICTDP1081; 2010-023026-20 (EudraCT Number)
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- NRT 60 (Experimental): A 6 mg dose of an experimental Nicotine Replacement Therapy (NRT) given every hour for 11 hours, with a 36-hour washout between visits
  Interventions: Drug: Nicotine
- NFG 60 (Active Comparator): A 4 mg dose of a marketed Nicotine Fruit Gum (NFG) given every hour for 11 hours, with a 36-hour washout between visits
  Interventions: Drug: Nicotine
- NRT 90 (Experimental): A 6 mg dose of NRT given every 90 minutes for 10.5 hours, with a 36-hour washout between visits
  Interventions: Drug: Nicotine
- NFG 90 (Active Comparator): A 4 mg dose of NFG given every 90 minutes for 10.5 hours, with a 36-hour washout between visits
  Interventions: Drug: Nicotine
- NIQ 60 (Active Comparator): A 4 mg dose of marketed nicotine mint lozenge (NIQ), given every hour for 11 hours, with a 36-hour washout between visits
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — 6 mg experimental Nicotine Replacement Therapy (NRT)
  Other Names: Not yet marketed
  Arms: NRT 60; NRT 90
Drug: Nicotine — 4 mg marketed Nicotine Fruit Gum (NFG)
  Other Names: Nicorette® Freshfruit Gum
  Arms: NFG 60; NFG 90
Drug: Nicotine — 4 mg marketed nicotine mint lozenge (NIQ)
  Other Names: NiQuitinTM Mint lozenge
  Arms: NIQ 60

SUMMARY:
Multiple-dose nicotine pharmacokinetics with three oral nicotine replacement products. A study in healthy smokers.

DETAILED DESCRIPTION:
Fifty (50) healthy male or female subjects between the ages of 19 and 50 years, inclusive, smoking at least 20 cigarettes daily during at least one year preceding inclusion. Multiple doses of all study treatments are given either every 60 minutes or every 90 minutes, respectively. All products will be administered in accordance with labeling, on five separate treatment visits. The subjects will abstain from smoking from 8 pm in the evening before and until the end of each visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, smoking at least 20 cigarettes daily during at least one year preceding inclusion.
* BMI between 17.5 and 30.0 kg/m2 and a total body weight of at least 55.0 kg.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.
* Willing and able to comply with all scheduled visits and study procedures

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.
* Any medical condition or history that might, per protocol or in the opinion of the investigator, compromise subject safety or trial results.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration | within the last dosing interval (starting at 10.5-11 hours after first product administration)
  Maximum Observed Plasma Concentration (Cmax), which is the maximum (peak) concentration (amount of drug) measurable in blood plasma within the last dosing interval, measured in nanograms/milliliter (ng/mL)
Average Concentration | within the last dosing interval (starting at 10.5-11 hours after first product administration)
  Average Nicotine Plasma Concentration (Cav) within the last dosing interval
Area Under the Curve | within the last dosing interval (starting at 10.5-11 hours after first product administration)
  Area under the nicotine plasma concentration-vs.-time curve during the last dosing interval (AUCt)

SECONDARY OUTCOMES:
Time of Maximum Concentration | During 12 hours post-dose
  The time at which maximum concentration is reached (Tmax)
Minimum Observed Concentration | within the last dosing interval (starting at 10.5-11 hours after first product administration)
  Minimum Observed Plasma Concentration (Cmin), which is the minimum concentration (amount of drug) measurable in blood plasma within the last dosing interval, measured in nanograms/milliliter (ng/mL)
Peak-Trough Fluctuation | within the last dosing interval (starting at 10.5-11 hours after first product administration)
  Percent of Peak-Trough Fluctuation in one dosing interval at steady state (PTF)
Swing | within the last dosing interval (starting at 10.5-11 hours after first product administration)
  Swing in one dosing interval at steady state, calculated as (Cmax-Cmin)/ Cmin
Nicotine Released | 30 minutes
  The amount of nicotine released from the product during product administration

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- McNeil AB Clinical Pharmacology R&D, Lund, Sweden